CLINICAL TRIAL: NCT03960866
Title: Randomized, Placebo-Controlled, Double-Masked Study of the Safety and Efficacy of Phentolamine Mesylate Ophthalmic Solution in Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy of Ophthalmic Phentolamine Mesylate in Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPI-NYXG-201 (ORION-1)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nyxol Ophthalmic Solution 1% (Experimental): 1 drop in each eye daily (QD) at or before bedtime (8pm to 10pm) for 14 days
  Interventions: Drug: Phentolamine Mesylate Ophthalmic Solution 1%
- Nyxol Ophthalmic Solution Vehicle (Placebo Comparator): 1 drop in each eye daily (QD) at or before bedtime (8pm to 10pm) for 14 days
  Interventions: Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo)

INTERVENTIONS:
Drug: Phentolamine Mesylate Ophthalmic Solution 1% — Topical Sterile Ophthalmic Solution
  Other Names: Nyxol®
  Arms: Nyxol Ophthalmic Solution 1%
Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo) — Topical Sterile Ophthalmic Solution
  Arms: Nyxol Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To evaluate the efficacy of Phentolamine Mesylate to lower intra-ocular pressure (IOP) in the treatment of Open-Angle Glaucoma (OAG) and Ocular Hypertension (OHT).
* To evaluate the ocular and systemic safety of Phentolamine Mesylate compared to its vehicle.
* To evaluate additional efficacy of Phentolamine Mesylate to improve visual performance.

DETAILED DESCRIPTION:
Placebo-controlled double-masked, multiple dose Phase 2 study in 40 patients with IOP ≥ 22 and ≤30 mmHg, evaluating ocular and systemic safety and efficacy following administration of Phentolamine mesylate 1.0% QD at 8PM to 10PM in both eyes for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT). A reported history of untreated OHT with IOP ≥22mmHg and ≤ 30mmHg is preferred.
3. Untreated or treated OAG/OHT with 2 or fewer ocular hypotensive medications.
4. Untreated (post-washout) mean IOP ≥ 22mmHg and ≤30mmHg in the study eye at the Qualification Visit (8AM).
5. Corrected visual acuity in each eye +1.0 logMAR or better by Early Treatment Diabetic Retinopathy Study (ETDRS) in each eye (equivalent to 20/200 or better) at the Screening Visit and Qualification Visit.
6. Otherwise healthy and well-controlled subjects.
7. Able and willing to give signed informed consent and follow study instructions.
8. Able to self-administer study medication or to have study medication administered by a caregiver throughout the study period.

Exclusion Criteria:

1. Closed or very narrow angles (Grade 0-1, Shaffer)
2. Glaucoma: pseudo-exfoliation or pigment dispersion component
3. Known hypersensitivity to any α-adrenoceptor antagonists
4. Previous laser and/or non-laser glaucoma surgery or procedure in either eye
5. Refractive surgery in either eye
6. Ocular trauma in either eye within the 6 months prior to Screening, or ocular surgery or non-refractive laser treatment within the 3 months prior to Screening
7. Recent or current evidence of ocular infection or inflammation in either eye
8. Ocular medication in either eye of any kind within 30 days of Screening
9. Clinically significant ocular disease in either eye
10. History of diabetic retinopathy
11. Contact lens wear within 3 days prior to and for the duration of the study
12. Central corneal thickness in either eye >600 μm at Screening
13. Any abnormality in either eye preventing reliable applanation tonometry
14. Known hypersensitivity or contraindication to α- and/or β-adrenoceptor antagonists
15. Clinically significant systemic disease that might interfere with the study
16. Participation in any investigational study within 30 days prior to Screening
17. Use of any topical or systemic adrenergic or cholinergic drugs up to 30 days prior to Screening, or during the study
18. Changes in systemic medication that could have an effect on IOP within 30 days prior to Screening
19. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control
20. Resting heart rate outside the normal range (50-110 beats per minute) at Screening or Qualification Visit
21. Hypertension with resting diastolic blood pressure (BP) > 105 mmHg or systolic BP > 160 mmHg at the Screening or Qualification Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - North Valley Eye Medical Group, Mission Hills, California
  - Clayton Eye Clinical Research, Morrow, Georgia
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Rochester Ophthalmological Group, Rochester, New York
  - Abrams Eye Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (13.23) | 63.2 (10.35) | 60.7 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 14 | 25
  Non-White | 8 | 6 | 14
Baseline Intraocular Pressure (Study Eye) [Mean (Standard Deviation); unit: mmHg] | 23.43 (1.675) | 24.38 (2.097) | 23.92 (1.939)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: change from Baseline in mean diurnal IOP in the study eye
Time Frame: 15 days
Population: Patients underwent a Screening visit where they were included in the trial if they were at least 18 years of age with either OHT in both eyes or OAG in 1 eye with OHT in the fellow eye, which was previously untreated or treated with ≤2 ocular hypotensive medications.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle
Number analyzed (Participants) | 18 | 19
mmHg | -2.30 (2.986) | -2.18 (1.856)
Statistical Analysis 1: Comparison: Nyxol Ophthalmic Solution 1% vs Nyxol Ophthalmic Solution Vehicle; Test type: Superiority; p = 0.89, t-test, 2 sided; Mean Difference (Net) = 0.12

2. Secondary Outcome: Pupil Diameter
Description: Change from Baseline Pupil Diameter (Photopic Conditions)
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle
Number analyzed (Participants) | 19 | 20
mm
  Day 8 (8AM) | -0.77 (0.538) | -0.07 (0.555)
  Day 15 (8AM) | -0.77 (0.550) | -0.01 (0.580)

3. Secondary Outcome: Distance Visual Acuity
Description: Percentage of Subjects Achieving ≥1 line improvement in Distance Visual Acuity from Baseline measured at 4 meters (photopic conditions)
Time Frame: 15 days
Population: Full Analysis Data Set
Measure: Count of Participants; unit: Participants
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle
Number analyzed (Participants) | 19 | 20
Participants | 12 | 4

4. Secondary Outcome: Conjunctival Hyperemia
Description: Conjunctival Hyperemia Category
Time Frame: 15 days
Population: Full analytical sample
Measure: Count of Participants; unit: Participants
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle
Number analyzed (Participants) | 19 | 20
Participants
  None | 4 | 8
  Mild | 10 | 8
  Moderate | 3 | 4
  Severe | 2 | 0

ADVERSE EVENTS:
Time Frame: 14 Days
Description: All treatment-emergent adverse events (TEAEs)/adverse reactions occurring during the study (ie, once the subject has received 1 dose of study medication) were documented, regardless of the assumption of causal relationship. All TEAEs/adverse reactions were documented from the time the subject received the first dose of study medication until the subject's participation in the study had completed.
Arm/Group | Nyxol Ophthalmic Solution 1% | Nyxol Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 5/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nyxol Ophthalmic Solution 1% (N=19) | Nyxol Ophthalmic Solution Vehicle (N=20)
Conjunctival Hyperemia (Eye disorders) | 3 | 1
Eye Pruritis (Eye disorders) | 1 | 0
Installation Site Discomfort (General disorders) | 3 | 0 — Installation Site Burning and/or Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03960866/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT03960866/SAP_003.pdf